CLINICAL TRIAL: NCT07344337
Title: Evaluation of the Effect of a Dietary Supplement Based on EGCG, Vitamin B12, Hyaluronic Acid, and Folic Acid on the Maintenance of Physiological Balance and the Natural Defenses of the Male Genital System in Subjects Exposed to HPV Infection.
Acronym: PERVI-I
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Lo.Li.Pharma s.r.l (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 8298
Record Dates: First submitted 2025-12-22; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: HPV Infection; Infertilities
Keywords: HPV; INFERTILITY
MeSH Terms: conditions — Papillomavirus Infections; Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients taking Pervistop (Experimental): 24 couples in which both partners will be treated with a combination of EGCG (200 mg), vitamin B12 (1 mg), hyaluronic acid (50 mg), and folic acid (400 µg), administered orally as one tablet once daily for 6 months.
  Interventions: Dietary Supplement: Pervistop
- Patients NO taking Pervistop (No Intervention): 24 couples who will not receive any supplementation

INTERVENTIONS:
Dietary Supplement: Pervistop — combination of EGCG, vitamin B12, hyaluronic acid, and folic acid.
  Arms: Patients taking Pervistop

SUMMARY:
This is a randomized pilot interventional study aimed at evaluating the effect of a dietary supplement containing EGCG, vitamin B12, hyaluronic acid, and folic acid on the maintenance of physiological balance and natural defenses of the male genital tract in subjects exposed to HPV infection and seeking care for infertility at natural procreation centers. The study includes 48 couples (96 participants) recruited at the International Scientific Institute "Paolo VI" of the A. Gemelli Policlinico, randomly assigned to two groups: 24 couples in which both partners receive one oral tablet per day of the supplement for 6 months, and 24 control couples receiving no supplementation. In addition to the primary objective, secondary outcomes assess potential support of sperm parameters, reproductive well-being of the couples, maintenance of genital mucosal physiological balance with possible reduction of HPV transmission risk to female partners, and support of physiological balance in the presence of co-infections or alterations of the genital microbiota.

DETAILED DESCRIPTION:
This randomized, pilot interventional study is designed to investigate the potential role of a dietary supplementation combining epigallocatechin gallate (EGCG), vitamin B12, hyaluronic acid, and folic acid in supporting the physiological balance and natural defense mechanisms of the male genital tract in subjects exposed to human papillomavirus (HPV) infection who are undergoing evaluation or treatment for infertility at natural procreation centers.

A total of 48 couples (96 participants) attending the outpatient clinics of the International Scientific Institute (ISI) "Paolo VI" at Policlinico A. Gemelli will be enrolled. All couples will include a male partner with documented HPV positivity. Participants will be randomly assigned, using a computer-generated randomization list, to one of two study arms. In the intervention group, 24 couples will receive an oral dietary supplement containing EGCG 200 mg, vitamin B12 1 mg, hyaluronic acid 50 mg, and folic acid 400 µg, administered as one tablet daily for a duration of six months to both partners. The control group will consist of 24 couples who will not receive any supplementation.

The primary objective of the study is to assess whether the combined supplementation contributes to the maintenance of physiological homeostasis and natural defense functions of the male genital system in individuals exposed to HPV. Secondary objectives include evaluating the potential effect of the supplementation on sperm quality parameters, the overall reproductive well-being of the couples, and the maintenance of genital mucosal physiological balance, with particular attention to factors that may influence the risk of HPV transmission to the female partner. Additionally, the study explores whether the supplementation supports physiological balance in the presence of possible co-infections or alterations of the genital microbiota.

As a pilot study, the results will provide preliminary data on feasibility, safety, and potential biological effects, contributing to the design of future larger-scale clinical investigations in this population.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Couple seeking pregnancy
* Male partner aged 25-65 years
* HPV DNA test indicating active HPV infection in the male partner
* HPV DNA test indicating negativity for HPV infection in the female partner

Exclusion Criteria:

* Concomitant diseases causing immunosuppression
* Treatment with immunomodulatory therapies
* Use of EGCG or other green tea extracts

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
The aim of the study is to evaluate the effect of a combination of EGCG, vitamin B12, hyaluronic acid, and folic acid on the maintenance of physiological balance and natural defense mechanisms of the male genital tract in subjects who, due to infertility | From enrollment to the end of treatment at 6 months
  The aim is to ensure continued HPV test negativity in the male partner throughout the six-month course of Pervistop therapy. The presence of the viral genotype will be determined by urethral swab sampling, followed by gene amplification using polymerase chain reaction (PCR) methodology.

CONTACTS AND LOCATIONS:
Overall Officials: Domenico Milardi, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ono A, Koshiyama M, Nakagawa M, Watanabe Y, Ikuta E, Seki K, Oowaki M. The Preventive Effect of Dietary Antioxidants on Cervical Cancer Development. Medicina (Kaunas). 2020 Nov 10;56(11):604. doi: 10.3390/medicina56110604. PMID 33182663
- [Background] Zhang D, Wen X, Wu W, Guo Y, Cui W. Elevated homocysteine level and folate deficiency associated with increased overall risk of carcinogenesis: meta-analysis of 83 case-control studies involving 35,758 individuals. PLoS One. 2015 May 18;10(5):e0123423. doi: 10.1371/journal.pone.0123423. eCollection 2015. PMID 25985325
- [Background] Ahn WS, Yoo J, Huh SW, Kim CK, Lee JM, Namkoong SE, Bae SM, Lee IP. Protective effects of green tea extracts (polyphenon E and EGCG) on human cervical lesions. Eur J Cancer Prev. 2003 Oct;12(5):383-90. doi: 10.1097/00008469-200310000-00007. PMID 14512803
- [Result] Weinberg M, Sar-Shalom Nahshon C, Feferkorn I, Bornstein J. Evaluation of human papilloma virus in semen as a risk factor for low sperm quality and poor in vitro fertilization outcomes: a systematic review and meta-analysis. Fertil Steril. 2020 May;113(5):955-969.e4. doi: 10.1016/j.fertnstert.2020.01.010. PMID 32386620
- [Result] Porcaro G, Pavone-Cossut MR, Moretti S, Bilotta G, Aragona C, Unfer V. Oral Treatment with EGCG, Folic Acid, Vitamin B12, and Hyaluronic Acid Improves HPV Clearance and Counteracts Its Persistence: A Clinical Study. Int J Mol Sci. 2025 May 29;26(11):5251. doi: 10.3390/ijms26115251. PMID 40508059
- [Result] Tinelli A, Gustapane S, Licchelli M, Coluccia AC, Panese G, Proietti S, Gambioli R. Treatment with Epigallocatechin Gallate, Folic Acid, Vitamin B12, and Hyaluronic Acid Decreases HPV Positivity in Women Attending Regional Screening in Puglia. Microorganisms. 2024 Sep 14;12(9):1897. doi: 10.3390/microorganisms12091897. PMID 39338571
- [Result] Aragona C, Bezerra Espinola MS, Bilotta G, Porcaro G, Calcagno M. Evaluating the Efficacy of Pervistop(R), a New Combination Based on EGCG, Folic Acid, Vitamin B12 and Hyaluronic Acid on Patients with Human Papilloma Virus (HPV) Persistent Infections and Cervical Lesions: A Pilot Study. J Clin Med. 2023 Mar 10;12(6):2171. doi: 10.3390/jcm12062171. PMID 36983172
- [Result] Kwanbunjan K., Saengkar P., Cheeramakara C., Thanomsak W., Benjachai W.,Laisupasin P., Buchachart K., Songmuaeng K., Boontaveeyuwat N. Low folate status as a risk factor for cervical dysplasia in Thai women. Nutr. Res. 2005;25:641-654. doi: 10.1016/j.nutres.2005.05.004.
- [Result] Hernandez BY, McDuffie K, Wilkens LR, Kamemoto L, Goodman MT. Diet and premalignant lesions of the cervix: evidence of a protective role for folate, riboflavin, thiamin, and vitamin B12. Cancer Causes Control. 2003 Nov;14(9):859-70. doi: 10.1023/b:caco.0000003841.54413.98. PMID 14682443
- [Result] Piyathilake CJ, Henao OL, Macaluso M, Cornwell PE, Meleth S, Heimburger DC, Partridge EE. Folate is associated with the natural history of high-risk human papillomaviruses. Cancer Res. 2004 Dec 1;64(23):8788-93. doi: 10.1158/0008-5472.CAN-04-2402. PMID 15574793
- [Result] Piyathilake CJ, Macaluso M, Chambers MM, Badiga S, Siddiqui NR, Bell WC, Edberg JC, Partridge EE, Alvarez RD, Johanning GL. Folate and vitamin B12 may play a critical role in lowering the HPV 16 methylation-associated risk of developing higher grades of CIN. Cancer Prev Res (Phila). 2014 Nov;7(11):1128-37. doi: 10.1158/1940-6207.CAPR-14-0143. Epub 2014 Aug 21. PMID 25145486
- [Result] Sedjo RL, Inserra P, Abrahamsen M, Harris RB, Roe DJ, Baldwin S, Giuliano AR. Human papillomavirus persistence and nutrients involved in the methylation pathway among a cohort of young women. Cancer Epidemiol Biomarkers Prev. 2002 Apr;11(4):353-9. PMID 11927495
- [Result] Yap JKW, Kehoe ST, Woodman CBJ, Dawson CW. The Major Constituent of Green Tea, Epigallocatechin-3-Gallate (EGCG), Inhibits the Growth of HPV18-Infected Keratinocytes by Stimulating Proteasomal Turnover of the E6 and E7 Oncoproteins. Pathogens. 2021 Apr 11;10(4):459. doi: 10.3390/pathogens10040459. PMID 33920477
- [Result] Zou C, Liu H, Feugang JM, Hao Z, Chow HH, Garcia F. Green tea compound in chemoprevention of cervical cancer. Int J Gynecol Cancer. 2010 May;20(4):617-24. doi: 10.1111/IGC.0b013e3181c7ca5c. PMID 20686382
- [Result] Chu C, Deng J, Man Y, Qu Y. Green Tea Extracts Epigallocatechin-3-gallate for Different Treatments. Biomed Res Int. 2017;2017:5615647. doi: 10.1155/2017/5615647. Epub 2017 Aug 13. PMID 28884125
- [Result] Tzellos TG, Sardeli C, Lallas A, Papazisis G, Chourdakis M, Kouvelas D. Efficacy, safety and tolerability of green tea catechins in the treatment of external anogenital warts: a systematic review and meta-analysis. J Eur Acad Dermatol Venereol. 2011 Mar;25(3):345-53. doi: 10.1111/j.1468-3083.2010.03796.x. PMID 21294779
- [Result] Tatti S, Swinehart JM, Thielert C, Tawfik H, Mescheder A, Beutner KR. Sinecatechins, a defined green tea extract, in the treatment of external anogenital warts: a randomized controlled trial. Obstet Gynecol. 2008 Jun;111(6):1371-9. doi: 10.1097/AOG.0b013e3181719b60. PMID 18515521
- [Result] Stockfleth E, Beti H, Orasan R, Grigorian F, Mescheder A, Tawfik H, Thielert C. Topical Polyphenon E in the treatment of external genital and perianal warts: a randomized controlled trial. Br J Dermatol. 2008 Jun;158(6):1329-38. doi: 10.1111/j.1365-2133.2008.08520.x. Epub 2008 Mar 20. PMID 18363746
- [Result] Gross G, Meyer KG, Pres H, Thielert C, Tawfik H, Mescheder A. A randomized, double-blind, four-arm parallel-group, placebo-controlled Phase II/III study to investigate the clinical efficacy of two galenic formulations of Polyphenon E in the treatment of external genital warts. J Eur Acad Dermatol Venereol. 2007 Nov;21(10):1404-12. doi: 10.1111/j.1468-3083.2007.02441.x. PMID 17958849
- [Result] Fiorillo L, Cervino G, Surace G, De Stefano R, Laino L, D'Amico C, Fiorillo MT, Meto A, Herford AS, Arzukanyan AV, Spagnuolo G, Cicciu M. Human Papilloma Virus: Current Knowledge and Focus on Oral Health. Biomed Res Int. 2021 Feb 1;2021:6631757. doi: 10.1155/2021/6631757. eCollection 2021. PMID 33623784
- [Result] Pal A, Kundu R. Human Papillomavirus E6 and E7: The Cervical Cancer Hallmarks and Targets for Therapy. Front Microbiol. 2020 Jan 21;10:3116. doi: 10.3389/fmicb.2019.03116. eCollection 2019. PMID 32038557
- [Result] Kato Y, Shigehara K, Nakagawa T, Nakata H, Iijima M, Nakashima K, Kawaguchi S, Izumi K, Kadono Y, Mizokami A. Human papillomavirus detected in sperm of Japanese infertile males affects reproductive parameters. Int J Infect Dis. 2021 Nov;112:294-299. doi: 10.1016/j.ijid.2021.09.029. Epub 2021 Sep 20. PMID 34547493
- [Result] Schillaci R, Capra G, Bellavia C, Ruvolo G, Scazzone C, Venezia R, Perino A. Detection of oncogenic human papillomavirus genotypes on spermatozoa from male partners of infertile couples. Fertil Steril. 2013 Nov;100(5):1236-40. doi: 10.1016/j.fertnstert.2013.06.042. Epub 2013 Jul 24. PMID 23891022
- [Result] De Toni L, Muscianisi F, Corsini C, Ghezzi M, Di Nisio A, Foresta C, Garolla A. Serum Anti-HPV Antibody Titer as a Marker of Vaccine Effectiveness in Males with Genital Infection. Vaccines (Basel). 2020 Dec 7;8(4):743. doi: 10.3390/vaccines8040743. PMID 33297367
- [Result] Foresta C, Noventa M, De Toni L, Gizzo S, Garolla A. HPV-DNA sperm infection and infertility: from a systematic literature review to a possible clinical management proposal. Andrology. 2015 Mar;3(2):163-73. doi: 10.1111/andr.284. Epub 2014 Oct 1. PMID 25270519
- [Result] Foresta C, Garolla A, Zuccarello D, Pizzol D, Moretti A, Barzon L, Palu G. Human papillomavirus found in sperm head of young adult males affects the progressive motility. Fertil Steril. 2010 Feb;93(3):802-6. doi: 10.1016/j.fertnstert.2008.10.050. Epub 2008 Dec 18. PMID 19100537
- [Result] Lenzi A, Mirone V, Gentile V, Bartoletti R, Ficarra V, Foresta C, Mariani L, Mazzoli S, Parisi SG, Perino A, Picardo M, Zotti CM. Rome Consensus Conference - statement; human papilloma virus diseases in males. BMC Public Health. 2013 Feb 7;13:117. doi: 10.1186/1471-2458-13-117. PMID 23391351
- [Result] Laprise C, Trottier H, Monnier P, Coutlee F, Mayrand MH. Prevalence of human papillomaviruses in semen: a systematic review and meta-analysis. Hum Reprod. 2014 Apr;29(4):640-51. doi: 10.1093/humrep/det453. Epub 2013 Dec 22. PMID 24365799
- [Result] Perez-Andino J, Buck CB, Ribbeck K. Adsorption of human papillomavirus 16 to live human sperm. PLoS One. 2009 Jun 9;4(6):e5847. doi: 10.1371/journal.pone.0005847. PMID 19513123
- [Result] Zacharis K, Messini CI, Anifandis G, Koukoulis G, Satra M, Daponte A. Human Papilloma Virus (HPV) and Fertilization: A Mini Review. Medicina (Kaunas). 2018 Jul 27;54(4):50. doi: 10.3390/medicina54040050. PMID 30344281
- [Result] Garolla A, Engl B, Pizzol D, Ghezzi M, Bertoldo A, Bottacin A, Noventa M, Foresta C. Spontaneous fertility and in vitro fertilization outcome: new evidence of human papillomavirus sperm infection. Fertil Steril. 2016 Jan;105(1):65-72.e1. doi: 10.1016/j.fertnstert.2015.09.018. Epub 2015 Oct 9. PMID 26453270
- [Result] Lorenzon L, Terrenato I, Dona MG, Ronchetti L, Rollo F, Marandino F, Carosi M, Diodoro MG, Sentinelli S, Visca P, Vocaturo G, Bellardini P, Vocaturo A, Benevolo M. Prevalence of HPV infection among clinically healthy Italian males and genotype concordance between stable sexual partners. J Clin Virol. 2014 Jul;60(3):264-9. doi: 10.1016/j.jcv.2014.04.003. Epub 2014 Apr 15. PMID 24794396
- [Result] Kero K, Rautava J. HPV Infections in Heterosexual Couples: Mechanisms and Covariates of Virus Transmission. Acta Cytol. 2019;63(2):143-147. doi: 10.1159/000494710. Epub 2019 Feb 22. PMID 30799413
- [Result] Widdice L, Ma Y, Jonte J, Farhat S, Breland D, Shiboski S, Moscicki AB. Concordance and transmission of human papillomavirus within heterosexual couples observed over short intervals. J Infect Dis. 2013 Apr 15;207(8):1286-94. doi: 10.1093/infdis/jit018. Epub 2013 Jan 14. PMID 23319742
- [Result] Giuliano AR, Nyitray AG, Kreimer AR, Pierce Campbell CM, Goodman MT, Sudenga SL, Monsonego J, Franceschi S. EUROGIN 2014 roadmap: differences in human papillomavirus infection natural history, transmission and human papillomavirus-related cancer incidence by gender and anatomic site of infection. Int J Cancer. 2015 Jun 15;136(12):2752-60. doi: 10.1002/ijc.29082. Epub 2014 Jul 26. PMID 25043222
- [Result] de Sanjose S, Serrano B, Castellsague X, Brotons M, Munoz J, Bruni L, Bosch FX. Human papillomavirus (HPV) and related cancers in the Global Alliance for Vaccines and Immunization (GAVI) countries. A WHO/ICO HPV Information Centre Report. Vaccine. 2012 Nov 20;30 Suppl 4:D1-83, vi. doi: 10.1016/S0264-410X(12)01435-1. No abstract available. PMID 23510764
- [Result] Doorbar J, Quint W, Banks L, Bravo IG, Stoler M, Broker TR, Stanley MA. The biology and life-cycle of human papillomaviruses. Vaccine. 2012 Nov 20;30 Suppl 5:F55-70. doi: 10.1016/j.vaccine.2012.06.083. PMID 23199966
- [Result] Cid Arregui A, Gariglio P, Kanda T, Doorbar J. ONCOGENIC HUMAN PAPILLOMAVIRUSES: High-Risk Human Papillomaviruses: Towards a Better Understanding of the Mechanisms of Viral Transformation, Latency and Immune-Escape. Open Virol J. 2012;6:160-2. doi: 10.2174/1874357901206010160. Epub 2012 Dec 28. No abstract available. PMID 23346264
- [Result] McLaughlin-Drubin ME, Munger K. Oncogenic activities of human papillomaviruses. Virus Res. 2009 Aug;143(2):195-208. doi: 10.1016/j.virusres.2009.06.008. Epub 2009 Jun 18. PMID 19540281
- [Result] Bosch FX, Broker TR, Forman D, Moscicki AB, Gillison ML, Doorbar J, Stern PL, Stanley M, Arbyn M, Poljak M, Cuzick J, Castle PE, Schiller JT, Markowitz LE, Fisher WA, Canfell K, Denny LA, Franco EL, Steben M, Kane MA, Schiffman M, Meijer CJ, Sankaranarayanan R, Castellsague X, Kim JJ, Brotons M, Alemany L, Albero G, Diaz M, de Sanjose S; ICO Monograph 'Comprehensive Control of HPV Infections and Related Diseases' Vaccine Volume 30, Supplement 5, 2012. Comprehensive control of human papillomavirus infections and related diseases. Vaccine. 2013 Dec 30;31 Suppl 6:G1-31. doi: 10.1016/j.vaccine.2013.10.002. PMID 24331817
- [Result] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338